CLINICAL TRIAL: NCT00809627
Title: A Prospective Trial of IV Caffeine vs Placebo for Post-Dural-Puncture Headache in the Emergency Department
Brief Title: Caffeine Versus Placebo for Spinal Headaches
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never initiated
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIP 2006 0051
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Post Dural Puncture Headache
Keywords: headache; caffeine; pain
MeSH Terms: conditions — Post-Dural Puncture Headache; Headache; Pain | interventions — Caffeine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): IV caffeine with saline and opiate
  Interventions: Drug: Caffeine
- 2 (Placebo Comparator): IV saline with opiate
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Caffeine — Caffeine 500 mg IV
  Other Names: Treatment group
  Arms: 1
Drug: saline — Normal saline
  Other Names: Placebo control group
  Arms: 2

SUMMARY:
Caffeine will be studied against placebo in patients with positional headache after a lumbar puncture (aka "spinal headache").

DETAILED DESCRIPTION:
Pain will be assessed at set intervals using a Visual Analog Scale. Blood patch therapy will be offered to all those still in pain at the end of one hour after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with post dural puncture headache

Exclusion Criteria:

* age < 18
* pregnant
* allergic to caffeine
* cardiac or peripheral vascular disease
* uncontrolled hypertension

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Pain as measured by Visual Analog Scale | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Kostic, MD, Study Chair — United States Naval Medical Center, Portsmouth; Marcelo Darabos, MD, Principal Investigator — United States Naval Medical Center, Portsmouth
Locations (1):
- Emergency Department, Naval Medical Center Portsmouth, Portsmouth, Virginia, United States